CLINICAL TRIAL: NCT00897988
Title: Effect of PI3K Inhibition in HPV-Associated HNSCC
Brief Title: DNA Analysis of Tumor Tissue Samples From Patients With Human Papilloma Virus-Associated Cancer of the Oropharynx
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000558955; P30CA068485 (NIH); VU-VICC-HN-0603; VU-VICC-IRB-060043
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Head and Neck Cancer
Keywords: recurrent squamous cell carcinoma of the oropharynx; stage I squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Gene Expression Profiling; Electrophoresis, Polyacrylamide Gel; Polymerase Chain Reaction; Reverse Transcriptase Polymerase Chain Reaction; Flow Cytometry; Immunoenzyme Techniques; Immunologic Techniques

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: mutation analysis
Genetic: polyacrylamide gel electrophoresis
Genetic: polymerase chain reaction
Genetic: protein expression analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: flow cytometry
Other: immunoenzyme technique
Other: immunologic technique
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Studying samples of tumor tissue in the laboratory from patients with cancer may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This laboratory study is looking at the DNA in tumor tissue samples from patients with human papilloma virus-associated cancer of the oropharynx.

DETAILED DESCRIPTION:
OBJECTIVES:

* Analyze PIK3CA expression and mutation and p110α amplification and expression in tumor tissue samples from patients with human papilloma virus positive (HPV+) and human papilloma virus negative (HPV-) squamous cell carcinoma (SCC) of the oropharynx.
* Determine proliferation and survival after PI3K inhibition in HPV(+) and HPV(-) oropharyngeal SCC cell lines and in HPV E6 and E7 expressing cells.
* Determine proliferation and survival after PI3K inhibition in short-term cultures of tumor tissue samples from patients with HPV(+) and HPV(-) primary SCC of the oropharynx.

OUTLINE: Previously collected tumor tissue samples are analyzed for HPV DNA by PCR amplification and direct sequencing of PCR products; expression of E6 protein and relative expression of PIK3CA by qRT-PCR; amplification of PIK3CA by Southern blotting; mutation of PIK3CA; expression of p110α, phospho-AKT, total AKT, and FOXO1 by polyacrylamide gel electrophoresis (PAGE) and immunoblotting; and the effect of PI3K inhibition on cell cycle and apoptosis by flow cytometry. Pharmacological studies are performed on oropharyngeal squamous cell carcinoma cell lines and short-term cultures and HPV E6 and E7 expressing cells using LY 294002 in vitro to analyze response to PI3K inhibition. Results of response to PI3K inhibition will be correlated with HPV status, PIK3CA expression, amplification, and mutation, and p110α expression.

PROJECTED ACCRUAL: A total of 20 HPV(+) and 20 HPV(-) tumor tissue specimens from patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Undergoing operative procedures for biopsy and/or resection of squamous cell carcinoma (SCC) of the oropharynx
* Tumor tissue sample available from the Head and Neck Tissue Repository and Clinical Database of Vanderbilt University
* No tumors with human papilloma virus (HPV) DNA sequences but no expression of E6

PATIENT CHARACTERISTICS:

* See Disease Characteristics

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-04

PRIMARY OUTCOMES:
PIK3CA expression and mutation and p110α amplification and expression in tumor tissue samples from patients with human papilloma virus positive (HPV+) and human papilloma virus negative (HPV-) squamous cell carcinoma (SCC) of the oropharynx
Proliferation and survival after PI3K inhibition in HPV(+) and HPV(-) oropharyngeal SCC cell lines and in HPV E6 and E7 expressing cells
Proliferation and survival after PI3K inhibition in short-term cultures of tumor tissues from patients with HPV(+) and HPV(-) primary SCC of the oropharynx

CONTACTS AND LOCATIONS:
Overall Officials: Wendell G. Yarbrough, MD, FACS, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee